CLINICAL TRIAL: NCT02298673
Title: Biomarker for Mucolipidosis Disorder Type I, II, III, IV AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGICAL PROTOCOL
Brief Title: Biomarker for Mucolipidosis Disorder Type I, II, III, IV (BioML)
Acronym: BioML
Status: Withdrawn | Type: Observational
Why Stopped: Transition into BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BML 06-2018
Record Dates: First submitted 2014-10-23; First posted 2014-11-24 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Skeletal Abnormalities; Psychomotor Retardation
Keywords: Mucolipidosis Disorder type I,II,III, IV; Biomarker
MeSH Terms: conditions — Psychomotor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectometry 10 ml EDTA blood or a dry blood spot filter card are taken. To proof the correct mucolipidosis disorder type I, II, III or IV diagnosis in those patients where up to the enrolment in the study no genetic testing has been done, sequencing of mucolipidosis disorder type I, II, III or IV will be done. The analyses will done in the Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with Mucolipidosis Disorder type I,II,III or IV or high-grade suspicion for Mucolipidosis Disorder type I,II,III or IV

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Mucolipidosis Disorder type I,II,III or IV from blood (plasma)

DETAILED DESCRIPTION:
Mucolipidoses (ML) are a group of inherited metabolic diseases in which both glycosaminoglycans (GAGs) and another group of substances called sphingolipids build up in the body. GAGs are long, repeating chains of complex sugar molecules, and sphingolipids are fats. ML disorders may also be referred to as "targeting defects" because affected individuals are lacking the enzyme (a protein that produces chemical reactions in the body) that "targets" other enzymes to the lysosome (a sac-like structure found in a cell).

Symptoms of ML can be congenital (present at birth) or begin in early childhood or adolescence. Early symptoms can include vision problems and developmental delays. Over time, many children with ML develop poor mental capacities, have difficulty reaching normal developmental milestones, and, in many cases, eventually die of the disease.

Changes in specific genes results in the deficiency or absence of the targeting enzyme. The ML disorders are categorized into four groups based on the clinical features and enzyme deficiencies. ML-II and ML-III are the more common forms of ML. An individual is usually suspected of having an ML disorder based on clinical features. The diagnosis is further confirmed by laboratory testing.

The mucolipidoses are inherited in an autosomal recessive manner, that is, they occur only when a child inherits two copies of the defective gene, one from each parent. When both parents carry a defective gene, each of their children faces a one in four chance of developing one of the MLs. At the same time, each child also faces a one in two chance of inheriting only one copy of the defective gene. People who have only one defective gene are known as carriers. These individuals do not develop the disease but they can pass the defective gene on to their own children. Because the defective genes involved in certain forms of ML are known, tests can identify people who are carriers in some instances.

The four types of ML are Sialidosis (sometimes referred to as ML I), and types II, III, and IV.

• Mucolipidosis type I (Sialidosis) The Sialidoses are autosomal recessive lysosomal storage disorders resulting from mutations in the NEU1 gene (6p21.3) which lead to an intracellular accumulation of glycoproteins containing sialic acid residues. Both types I and II are caused by mutations in the same gene.

ML1 (NEU1 deficiency) is a neurodegenerative disorder with progressive deterioration of muscle and central nervous system functions. Myoclonus, mental deterioration, hepatosplenomegaly, muscle weakness and atrophy are common. The defect in neuraminidase activity leads to abnormal amounts of sialyl-oligosaccharides in the urine. Spinal deformities such as kyphosis are common. Deep tendon reflexes are exaggerated. Ataxia and hearing loss may be present. Coarse facies, a barrel chest, and short stature are characteristic. Hepatic cells contain numerous vacuoles and numerous inclusions.

A cherry red spot is may be seen in late childhood or early adolescence. It occurs in nearly 100% of patients with type I while only 75% of type II patients have this feature possibly because their early death from the more severe systemic disease prevents full ascertainment. Visual acuity is reduced, sometimes severely. Some but not all individuals have corneal and lens opacities. A subtle corneal haze has also been seen. Nystagmus has been reported.

Sialidosis types I and II are both caused by mutations in the neuraminidase gene. Type I is associated with milder disease than type II which has an earlier age of onset and may present in infancy or even begin in utero. Early death within two years of age is common in the congenital or infantile forms. There is, however, significant variability in age of onset and the course of disease among types.

• Mucolipidosis type II (I-Cell Disease) I-cell disease (mucolipidosis II) is a rare inherited metabolic disorder characterized by coarse facial features, skeletal abnormalities and mental retardation. The symptoms of I-cell disease are similar to but more severe than those of Hurler syndrome. The symptoms associated with this disorder typically become obvious during infancy and may include multiple abnormalities of the skull and face and growth delays.

This disorder belongs to a group of diseases known as lysosomal storage disorders. Lysosomes are particles bound in membranes within cells that break down certain fats and carbohydrates. Multiple enzyme deficiencies associated with I-cell disease lead to the accumulation of certain fatty substances (mucolipids) and certain complex carbohydrates (mucopolysaccharides) within the cells of many tissues of the body.

I-cell disease is caused by a mutation in the GNPTAB gene that leads to a deficiency in the enzyme UDP-N-acetylglucoseamine-1-phosphotransferase. I-cell disease is inherited as an autosomal recessive genetic trait.

• Mucolipidosis type III (Pseudo-Hurler Polydystrophy) Mucolipidosis III alpha/beta is a slowly progressive disorder that affects many parts of the body. Signs and symptoms of this condition typically appear around age 3.

Individuals with mucolipidosis III alpha/beta grow slowly and have short stature. They also have stiff joints and dysostosis multiplex, which refers to multiple skeletal abnormalities seen on x-ray. Many affected individuals develop low bone mineral density (osteoporosis), which weakens the bones and makes them prone to fracture. Osteoporosis and progressive joint problems also cause pain in people with mucolipidosis III alpha/beta, which becomes more severe over time.

People with mucolipidosis III alpha/beta often have heart valve abnormalities and mild clouding of the clear covering of the eye (cornea). Their facial features become slightly thickened or "coarse" over time. Affected individuals may also develop frequent ear and respiratory infections. About half of people with this condition have mild intellectual disability or learning problems. Individuals with mucolipidosis III alpha/beta generally survive into adulthood, but they may have a shortened lifespan.

Mucolipidosis III alpha/beta is a rare disorder, although its exact prevalence is unknown. It is estimated to occur in about 1 in 100,000 to 400,000 individuals worldwide Mutations in the GNPTAB gene cause mucolipidosis III alpha/beta. This gene provides instructions for making a part (subunit) of an enzyme called GlcNAc-1-phosphotransferase. This enzyme helps prepare certain newly made enzymes for transport to lysosomes. Lysosomes are compartments within the cell that use digestive enzymes to break down large molecules into smaller ones that can be reused by cells. GlcNAc-1-phosphotransferase is involved in the process of attaching a molecule called mannose-6-phosphate (M6P) to specific digestive enzymes. Just as luggage is tagged at the airport to direct it to the correct destination, enzymes are often "tagged" after they are made so they get to where they are needed in the cell. M6P acts as a tag that indicates a digestive enzyme should be transported to the lysosome.

Mutations in the GNPTAB gene that cause mucolipidosis III alpha/beta result in reduced activity of GlcNAc-1-phosphotransferase. These mutations disrupt the tagging of digestive enzymes with M6P, which prevents many enzymes from reaching the lysosomes. Digestive enzymes that do not receive the M6P tag end up outside the cell, where they have increased activity. The shortage of digestive enzymes within lysosomes causes large molecules to accumulate. Conditions that cause molecules to build up inside lysosomes, including mucolipidosis III alpha/beta, are called lysosomal storage disorders. The signs and symptoms of mucolipidosis III alpha/beta are most likely due to the shortage of digestive enzymes inside lysosomes and the effects these enzymes have outside the cell.

Mutations in the GNPTAB gene can also cause a similar but more severe disorder called mucolipidosis II alpha/beta. These mutations completely eliminate the function of GlcNAc-1-phosphotransferase. Mucolipidosis III alpha/beta and mucolipidosis II alpha/beta represent two ends of a spectrum of disease severity.

• Mucolipidosis type IV Mucolipidosis type IV (caused by mutations in the MCOLN1 gene) is an inherited disorder characterized by delayed development and progressive vision loss. The severe form of the disorder is called typical mucolipidosis type IV, and the mild form is called atypical mucolipidosis type IV.

Approximately 95 percent of individuals with this condition have the severe form. People with typical mucolipidosis type IV have delayed development of mental and motor skills (psychomotor delay). Motor skills including: sitting, standing, walking, grasping objects, and writing. Psychomotor delay is moderate to severe and usually becomes apparent during the first year of life. Affected individuals have intellectual disability, limited or absent speech, difficulty chewing and swallowing, weak muscle tone (hypotonia) that gradually turns into abnormal muscle stiffness (spasticity), and problems controlling hand movements. Most people with typical mucolipidosis type IV are unable to walk independently. In about 15 percent of affected individuals, the psychomotor problems worsen over time.

Vision may be normal at birth in people with typical mucolipidosis type IV, but it becomes increasingly impaired during the first decade of life. Individuals with this condition develop clouding of the clear covering of the eye (cornea) and progressive breakdown of the light-sensitive layer at the back of the eye (retina). By their early teens, affected individuals have severe vision loss or blindness.

People with typical mucolipidosis type IV also have impaired production of stomach acid (achlorhydria). Achlorhydria does not cause any symptoms in these individuals, but it does result in unusually high levels of gastrin in the blood. Gastrin is a hormone that regulates the production of stomach acid. Individuals with mucolipidosis type IV may not have enough iron in their blood, which can lead to a shortage of red blood cells (anemia). People with the severe form of this disorder usually survive to adulthood; however, they may have a shortened lifespan.

About 5 percent of affected individuals have atypical mucolipidosis type IV. These individuals usually have mild psychomotor delay and may develop the ability to walk. People with atypical mucolipidosis type IV tend to have milder eye abnormalities than those with the severe form of the disorder. Achlorhydria also may be present in mildly affected individuals.

Mucolipidosis type IV is estimated to occur in 1 in 40,000 people. About 70 percent of affected individuals have Ashkenazi Jewish ancestry.

Mutations in the MCOLN1 gene cause mucolipidosis type IV. This gene provides instructions for making a protein called mucolipin-1. This protein is located in the membranes of lysosomes and endosomes, compartments within the cell that digest and recycle materials. While its function is not completely understood, mucolipin-1 plays a role in the transport (trafficking) of fats (lipids) and proteins between lysosomes and endosomes. Mucolipin-1 appears to be important for the development and maintenance of the brain and retina. In addition, this protein is likely critical for normal functioning of the cells in the stomach that produce digestive acids.

Most mutations in the MCOLN1 gene result in the production of a non-functional protein or prevent any protein from being produced. A lack of functional mucolipin-1 impairs transport of lipids and proteins, causing these substances to build up inside lysosomes. Conditions that cause molecules to accumulate inside the lysosomes, including mucolipidosis type IV, are called lysosomal storage disorders. Two mutations in the MCOLN1 gene account for almost all cases of mucolipidosis type IV in people with Ashkenazi Jewish ancestry. It remains unclear how mutations in this gene lead to the signs and symptoms of mucolipidosis type IV.

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood (plasma) of affected patients that allow diagnosing in the future the Disorder earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to identify and validate a new biochemical marker from the plasma of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment. Examining blood samples will allow determining whether measurement is feasible in blood samples and will further promote early detection of mucolipidosis disorder type I, II, III or IV.

ELIGIBILITY:
INCLUSION CRITERIA

* Informed consent will be obtained from the parents before any study related procedures.
* Patients of both genders older than 2 month
* The patient has a diagnosis of Mucolipidosis Disorder type I,II,III or IV or high-grade suspicion for Mucolipidosis Disorder type I,II,III or IV
* High-grade suspicion present, if one or more inclusion criteria are valid:

Positive family anamnesis for Mucolipidosis Disorder type I,II,III or IV

Skeletal abnormalities

Psychomotor retardation

Progressive failure to thrive

Hoarse voice

EXCLUSION CRITERIA

* No Informed consent from the parents before any study related procedures.
* Patients of both genders younger than 2 month
* No diagnosis of Mucolipidosis Disorder type I,II,III or IV or no valid criteria for profound suspicion of Mucolipidosis Disorder type I,II,III or IV

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Mucolipidosis Disorder type I,II,III or IV or high-grade suspicion for Mucolipidosis Disorder type I,II,III or IV
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Mucolipidosis disorder type I, II, III or IV from blood (plasma). | 12 months

SECONDARY OUTCOMES:
Testing for clinical robustness, specificity and long-term stability of the biomarker. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (5):
- Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt
- Centogene AG, Rostock, Germany
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - NIRMAN-University of Mumbai-Institute of Research in Mental and Neurological handicap, Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided